CLINICAL TRIAL: NCT01045421
Title: A Phase 1 Dose Escalation Study of MLN8237, an Aurora A Kinase Inhibitor, in Adult Patients With Nonhematological Malignancies, Followed by a Phase 2 of MLN8237 in Lung, Breast, Head and Neck, or Gastroesophageal Malignancies
Brief Title: Alisertib in Adults With Nonhematological Malignancies, Followed by Alisertib in Lung, Breast, Head and Neck or Gastroesophageal Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C14007; 2008-006981-27 (EudraCT Number); U1111-1171-0859 (Registry Identifier: WHO)
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-07

CONDITIONS: Advanced Nonhematological Malignancies; Non-Small Cell Lung Cancer; Small Cell Lung Cancer; Metastatic Breast Cancer; Head and Neck Squamous Cell Carcinoma; Gastroesophageal Adenocarcinoma
Keywords: NSCLC; SCLC; HNSCC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MLN8237 (Alisertib) (Experimental): MLN8237 administered as an enteric-coated tablet (ECT)
  Interventions: Drug: MLN8237 (Alisertib)

INTERVENTIONS:
Drug: MLN8237 (Alisertib) — Phase 1:
  MLN8237 will be administered orally twice a day on a 7-day dosing schedule
  Phase 2:
  MLN8237 will be administered orally at the maximum tolerated dose determined in Phase 1 for 7-days followed by a minimum 14-day rest period.

SUMMARY:
This is an open-label, multicenter study with a phase 1 dose escalation portion and a 2-stage, phase 2 portion, investigating MLN8237 (alisertib) in patients with advanced nonhematological malignancies.

DETAILED DESCRIPTION:
Following the determination of the Recommended Phase 2 Dose (RP2D) and schedule (Phase 1), 20 response-evaluable patients in each of the 5 tumor indications will be enrolled (Phase 2-Stage 1). An interim analysis will determine which tumor indications will proceed to enroll an additional 25 patients (Phase 2-Stage 2) to further evaluate Overall Response Rate (ORR) and other secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* 18 years or older
* Histologically or cytologically confirmed metastatic and/or advanced solid tumor (Phase 1 only)
* Phase 2 requires Non-small cell lung cancer (NSCLC); Small-cell lung cancer; Breast adenocarcinoma (female patients only); Squamous cell cancer of the head and neck (HNSCC); or Gastroesophageal adenocarcinoma
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Female patients who are post menopausal, surgically sterile, or agree to practice 2 effective methods of contraception or abstain from heterosexual intercourse
* Male patients who agree to practice effective barrier contraception or agree to abstain from heterosexual intercourse
* Voluntary written consent
* Wiling to comply with scheduled visits, treatment plan, laboratory tests and other trial procedures
* Measurable disease (Phase 2 only)

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

* Female patients who are pregnant or lactating
* Serious medical or psychiatric illness that could interfere with protocol completion
* Receipt of more than 2 previous cytotoxic chemotherapeutic regimens (4 previous regimens for breast cancer). There is no limit on the number of prior noncytotoxic therapies
* Prior treatment with Aurora A-targeted agents, including MLN8237
* Prior treatment with high-dose chemotherapy
* Prior allogeneic bone marrow or other organ transplant
* Antineoplastic therapy, radiation therapy or any experimental therapy 21 days prior to first dose of MLN8237
* Symptomatic brain metastasis
* Radiotherapy to greater than 25% of bone marrow
* Diagnosis or treatment of another malignancy within 2 years preceding first dose of study drug except nonmelanoma skin cancer or in situ malignancy completely resected
* Myocardial infarction within 6 months of enrollment
* Uncontrolled cardiovascular condition
* Major surgery within 14 days of first dose of MLN8237
* Active infection requiring systemic therapy, or other serious infection
* Inability to swallow oral medication
* Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C
* Patients requiring full systemic anticoagulation
* History of uncontrolled sleep apnea syndrome
* Treatment with clinically significant enzyme inducers within 14 days prior to the first dose of MLN8237 and during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2010-02; Primary Completion 2013-05 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (2):
- United States (2):
  - Houston, Texas
  - Salt Lake City, Utah

REFERENCES:
- [Derived] Melichar B, Adenis A, Lockhart AC, Bennouna J, Dees EC, Kayaleh O, Obermannova R, DeMichele A, Zatloukal P, Zhang B, Ullmann CD, Schusterbauer C. Safety and activity of alisertib, an investigational aurora kinase A inhibitor, in patients with breast cancer, small-cell lung cancer, non-small-cell lung cancer, head and neck squamous-cell carcinoma, and gastro-oesophageal adenocarcinoma: a five-arm phase 2 study. Lancet Oncol. 2015 Apr;16(4):395-405. doi: 10.1016/S1470-2045(15)70051-3. Epub 2015 Feb 27. PMID 25728526
- [Derived] Falchook G, Kurzrock R, Gouw L, Hong D, McGregor KA, Zhou X, Shi H, Fingert H, Sharma S. Investigational Aurora A kinase inhibitor alisertib (MLN8237) as an enteric-coated tablet formulation in non-hematologic malignancies: phase 1 dose-escalation study. Invest New Drugs. 2014 Dec;32(6):1181-7. doi: 10.1007/s10637-014-0121-6. Epub 2014 Jun 1. PMID 24879333

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 42 investigative sites in France, Poland, the Czech Republic, and the United States from 16 February 2010 to 25 April 2014.
Pre-assignment Details: Participants with a historical diagnosis of relapsed or refractory advanced nonhematological malignancies were enrolled in 1 of the 2 stages, Phase 1 (lead-in alisertib dose escalation stage) and Phase 2 (efficacy and safety assessment stage for alisertib dose determined in Phase 1).
Groups:
- Phase 1: MLN8237 10 mg: MLN8237 (alisertib) 10 milligram (mg), enteric-coated tablets, orally, twice daily for 7 days followed by 14 days of rest period in 21-day treatment cycles for a maximum of 24 months, or until progressive disease, unacceptable treatment-related toxicity, or initiation of a different anticancer therapy during Phase 1 portion of the study.
- Phase 1: MLN8237 20 mg: MLN8237 (alisertib) 20 mg, enteric-coated tablets, orally, twice daily for 7 days followed by 14 days of rest period in 21-day treatment cycles for a maximum of 24 months, or until progressive disease, unacceptable treatment-related toxicity, or initiation of a different anticancer therapy during Phase 1 portion of the study.
- Phase 1: MLN8237 40 mg: MLN8237 (alisertib) 40 mg, enteric-coated tablets, orally, twice daily for 7 days followed by 14 days of rest period in 21-day treatment cycles for a maximum of 24 months, or until progressive disease, unacceptable treatment-related toxicity, or initiation of a different anticancer therapy during Phase 1 portion of the study.
- Phase 1: MLN8237 50 mg: MLN8237 (alisertib) 50 mg, enteric-coated tablets, orally, twice daily for 7 days followed by 14 days of rest period in 21-day treatment cycles for a maximum of 24 months, or until progressive disease, unacceptable treatment-related toxicity, or initiation of a different anticancer therapy during Phase 1 portion of the study.
- Phase 1: MLN8237 60 mg: MLN8237 (alisertib) 60 mg, enteric-coated tablets, orally, twice daily for 7 days followed by 14 days of rest period in 21-day treatment cycles for a maximum of 24 months, or until progressive disease, unacceptable treatment-related toxicity, or initiation of a different anticancer therapy during Phase 1 portion of the study.
- Phase 1: MLN8237 50 mg- Pancreatic Cancer: MLN8237 (alisertib) 50 mg, enteric-coated tablets, orally, twice daily for 7 days followed by 14 days of rest period in 21-day treatment cycles for a maximum of 24 months, or until progressive disease, unacceptable treatment-related toxicity, or initiation of a different anticancer therapy in participants with pancreatic cancer during Phase 1 portion of the study.
- Phase 2: MLN8237 50 mg- Breast Cancer: MLN8237 (alisertib) 50 mg, enteric-coated tablets, orally, twice daily for 7 days followed by 14 days of rest period in 21-day treatment cycles for a maximum of 24 months, or until progressive disease, unacceptable treatment-related toxicity, or initiation of a different anticancer therapy in participants with breast cancer during Phase 2 portion of the study.
- Phase 2: MLN8237 50 mg- Gastric Cancer: MLN8237 (alisertib) 50 mg, enteric-coated tablets, orally, twice daily for 7 days followed by 14 days of rest period in 21-day treatment cycles for a maximum of 24 months, or until progressive disease, unacceptable treatment-related toxicity, or initiation of a different anticancer therapy in participants with gastric cancer during Phase 2 portion of the study.
- Phase 2: MLN8237 50 mg- HNSCC: MLN8237 (alisertib) 50 mg, enteric-coated tablets, orally, twice daily for 7 days followed by 14 days of rest period in 21-day treatment cycles for a maximum of 24 months, or until progressive disease, unacceptable treatment-related toxicity, or initiation of a different anticancer therapy in participants with head and neck squamous cell carcinoma (HNSCC) during Phase 2 portion of the study.
- Phase 2: MLN8237 50 mg- NSCLC: MLN8237 (alisertib) 50 mg, enteric-coated tablets, orally, twice daily for 7 days followed by 14 days of rest period in 21-day treatment cycles for a maximum of 24 months, or until progressive disease, unacceptable treatment-related toxicity, or initiation of a different anticancer therapy in participants with non-small cell lung cancer (NSCLC) during Phase 2 portion of the study.
- Phase 2: MLN8237 50 mg- SCLC: MLN8237 (alisertib) 50 mg, enteric-coated tablets, orally, twice daily for 7 days followed by 14 days of rest period in 21-day treatment cycles for a maximum of 24 months, or until progressive disease, unacceptable treatment-related toxicity, or initiation of a different anticancer therapy in participants with small cell lung cancer (SCLC) during Phase 2 portion of the study.
Period: Phase 1
Arm/Group | Phase 1: MLN8237 10 mg | Phase 1: MLN8237 20 mg | Phase 1: MLN8237 40 mg | Phase 1: MLN8237 50 mg | Phase 1: MLN8237 60 mg | Phase 1: MLN8237 50 mg- Pancreatic Cancer | Phase 2: MLN8237 50 mg- Breast Cancer | Phase 2: MLN8237 50 mg- Gastric Cancer | Phase 2: MLN8237 50 mg- HNSCC | Phase 2: MLN8237 50 mg- NSCLC | Phase 2: MLN8237 50 mg- SCLC
Started | 1 | 3 | 4 | 12 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 3 | 4 | 11 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1: MLN8237 10 mg | Phase 1: MLN8237 20 mg | Phase 1: MLN8237 40 mg | Phase 1: MLN8237 50 mg | Phase 1: MLN8237 60 mg | Phase 1: MLN8237 50 mg- Pancreatic Cancer | Phase 2: MLN8237 50 mg- Breast Cancer | Phase 2: MLN8237 50 mg- Gastric Cancer | Phase 2: MLN8237 50 mg- HNSCC | Phase 2: MLN8237 50 mg- NSCLC | Phase 2: MLN8237 50 mg- SCLC
Started | 0 | 0 | 0 | 0 | 0 | 0 | 53 | 55 | 55 | 26 | 60
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 53 | 50 | 53 | 23 | 58
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 3 | 2
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: MLN8237- All Participants: MLN8237 (alisertib) 10, 20, 30, 40, 50, or 60 mg enteric-coated tablets, orally, twice daily, for 7 days followed by 14 days of rest period in 21-day treatment cycles for a maximum of 24 months, or until progressive disease, unacceptable treatment-related toxicity, or initiation of a different anticancer therapy in participants enrolled in dose-escalation or pancreatic cancer cohort during Phase 1 portion of the study.
- Total: Total of all reporting groups
Arm/Group | Phase 1: MLN8237- All Participants | Phase 2: MLN8237 50 mg- Breast Cancer | Phase 2: MLN8237 50 mg- Gastric Cancer | Phase 2: MLN8237 50 mg- HNSCC | Phase 2: MLN8237 50 mg- NSCLC | Phase 2: MLN8237 50 mg- SCLC | Total
Number analyzed (Participants) | 24 | 53 | 55 | 55 | 26 | 60 | 273
Age, Customized [Number; unit: participants]
  18-64 years | 17 | 37 | 33 | 38 | 17 | 38 | 180
  65-84 years | 7 | 16 | 21 | 17 | 9 | 22 | 92
  85 years and over | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 53 | 12 | 3 | 12 | 28 | 117
  Male | 15 | 0 | 43 | 52 | 14 | 32 | 156
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 3 | 4 | 2 | 1 | 1 | 1 | 12
  Not Hispanic or Latino | 19 | 48 | 49 | 50 | 25 | 57 | 248
  Not reported | 2 | 1 | 4 | 4 | 0 | 2 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  White | 18 | 49 | 51 | 53 | 22 | 56 | 249
  Black or African American | 3 | 1 | 3 | 2 | 2 | 4 | 15
  Asian | 2 | 1 | 0 | 0 | 1 | 0 | 4
  Chinese | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Other | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Not reported | 1 | 1 | 1 | 0 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  Czech Republic | 0 | 19 | 20 | 8 | 7 | 15 | 69
  France | 0 | 10 | 8 | 11 | 3 | 8 | 40
  Poland | 0 | 1 | 0 | 1 | 0 | 7 | 9
  United States | 24 | 23 | 27 | 35 | 16 | 30 | 155
Disease stage at study entry [Number; unit: participants] — Assessment of disease stage for Medical History and Physical Examination at baseline were assessed according to the criteria set by the American Joint Committee on Cancer Tumor Staging version 7.0. The exact definition of a stage vary depending on the tumor type. Stage I cancers are the least advanced and often have a better prognosis. Higher stage cancers are often more advanced but in many cases can still be treated successfully.
  participants
    IA | 1 | 0 | 0 | 0 | 0 | 0 | 1
    II | 0 | 0 | 0 | 1 | 0 | 0 | 1
    III | 1 | 0 | 1 | 2 | 0 | 0 | 4
    IIIA | 1 | 1 | 0 | 0 | 0 | 1 | 3
    IIIB | 0 | 3 | 0 | 0 | 5 | 2 | 10
    IIIC | 0 | 1 | 0 | 0 | 0 | 0 | 1
    IV | 19 | 48 | 54 | 2 | 21 | 57 | 201
    IVA | 1 | 0 | 0 | 23 | 0 | 0 | 24
    IVB | 1 | 0 | 0 | 2 | 0 | 0 | 3
    IVC | 0 | 0 | 0 | 25 | 0 | 0 | 25
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: participants] — ECOG performance status assesses a participant's physical ability on a 6-point scale: 0=fully active, able to carry on all predisease activities without restriction; 1=restricted in physically strenuous activity, ambulatory and able to carry out light or sedentary work; 2=ambulatory (>50% of waking hours), capable of all self care, unable to carry out any work activities; 3=capable of only limited self care, confined to bed/chair >50% of waking hours; 4=completely disabled, cannot carry on any self care, totally confined to bed/chair; 5=dead.
  participants
    0 | 4 | 23 | 21 | 17 | 7 | 13 | 85
    1 | 20 | 30 | 34 | 38 | 19 | 47 | 188

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: Toxicity according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0. DLT defined as any of the following considered related to alisertib by investigator: Grade 4 neutropenia (absolute neutrophil count <500 cells/cubic meter [cells/mm^3]) for >7 days; Grade 4 neutropenia with coincident fever; Grade 4 thrombocytopenia (platelets <25,000 cells/mm3) for >7 days; Platelet count <10,000 cells/mm3; Grade 3 thrombocytopenia with clinically significant bleeding; Delay in initiation of the subsequent therapy cycle by >7 days due to treatment-related toxicity; >=Grade 3 nonhematological toxicity except >=Grade 3 nausea/emesis occurred in the absence of optimal antiemetic therapy; >=Grade 3 diarrhea occurred in the absence of optimal supportive therapy with loperamide/comparable antidiarrheal; Grade 3 fatigue for <1 week; Other Grade 3 nonhematological toxicity that could be safely, reliably controlled to <=Grade 2 with appropriate treatment.
Time Frame: Phase 1: Cycle 1 Day 1 to Cycle 2 Day 21
Population: DLT-Evaluable population: all participants in the Phase 1 portion of the study who either experienced DLT during Cycle 1 or completed at least 85% of the planned doses of alisertib and had sufficient follow-up data to allow the investigators and sponsor to determine whether DLT occurred.
Measure: Number; unit: participants
Arm/Group | Phase 1: MLN8237 10 mg | Phase 1: MLN8237 20 mg | Phase 1: MLN8237 40 mg | Phase 1: MLN8237 50 mg | Phase 1: MLN8237 60 mg | Phase 1: MLN8237 50 mg- Pancreatic Cancer
Number analyzed (Participants) | 1 | 3 | 4 | 12 | 3 | 1
participants | 0 | 0 | 0 | 2 | 0 | 0

2. Primary Outcome: Phase 2: Percentage of Participants With Objective Response
Description: Percentage of participants with objective response based assessment of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST). CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis less than [<] 10 millimeter [mm]). No new lesions. PR was defined as greater than or equal to (>=) 30 percent (%) decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: Baseline until complete response or partial response, assessed every 2 cycles up to end of study (up to 50 cycles)
Population: Response-Evaluable population included all participants with measurable disease who received at least 1 dose of alisertib and had at least 1 post-baseline response assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: MLN8237 50 mg- Breast Cancer | Phase 2: MLN8237 50 mg- Gastric Cancer | Phase 2: MLN8237 50 mg- HNSCC | Phase 2: MLN8237 50 mg- NSCLC | Phase 2: MLN8237 50 mg- SCLC
Number analyzed (Participants) | 49 | 47 | 45 | 23 | 48
percentage of participants | 18 [9 to 32] | 9 [2 to 20] | 9 [2 to 21] | 4 [0 to 22] | 21 [10 to 35]

3. Secondary Outcome: Phase 2: Progression-free Survival (PFS)
Description: PFS was defined as the time from randomization (or the first dose of study treatment for non-randomized studies) to the first documentation of objective tumor progression or to death due to any cause, whichever occurred first. Tumor progression as per RECIST 1.1 was defined as at least 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of 1or more new lesions is also considered progression.
Time Frame: Baseline until progressive disease, assessed every 2 cycles up to end of study (up to 50 cycles)
Population: Safety population included all participants who received any amount of alisertib.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 2: MLN8237 50 mg- Breast Cancer | Phase 2: MLN8237 50 mg- Gastric Cancer | Phase 2: MLN8237 50 mg- HNSCC | Phase 2: MLN8237 50 mg- NSCLC | Phase 2: MLN8237 50 mg- SCLC
Number analyzed (Participants) | 53 | 55 | 55 | 26 | 60
days | 164 [78 to 239] | 49 [41 to 78] | 72 [43 to 96] | 92 [72 to 120] | 49 [42 to 96]

4. Secondary Outcome: Phase 2: Time to Disease Progression (TTP)
Description: Time in days from start of study treatment to first documentation of objective tumor progression. Tumor progression as per RECIST 1.1 was defined as at least 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of 1or more new lesions is also considered progression.
Time Frame: Baseline until disease progression, assessed every 2 cycles up to end of study (up to 50 cycles)
Population: Safety population included all participants who received any amount of alisertib.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 2: MLN8237 50 mg- Breast Cancer | Phase 2: MLN8237 50 mg- Gastric Cancer | Phase 2: MLN8237 50 mg- HNSCC | Phase 2: MLN8237 50 mg- NSCLC | Phase 2: MLN8237 50 mg- SCLC
Number analyzed (Participants) | 53 | 55 | 55 | 26 | 60
days | 164 [78 to 239] | 46 [40 to 86] | 72 [43 to 96] | 92 [74 to 144] | 78 [42 to 114]

5. Secondary Outcome: Phase 2: Duration of Response (DOR)
Description: Time in days from the first documentation of objective tumor response to objective tumor progression or death due to any cancer. Duration of tumor response=(the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1). CR: complete disappearance of all target lesions and non-target disease, except nodal disease; all nodes decreased to normal; no new lesions. PR: >=30% decrease under baseline of the sum of diameters of all target lesions; no unequivocal progression of non-target disease; no new lesions. Tumor progression: >=20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study); absolute increase of >=5 mm; appearance of >=1 new lesions is also considered progression. DOR calculated for the subgroup of participants with objective response.
Time Frame: Baseline up to Week 50
Population: Included a subset of response-evaluable population who had objective tumor response.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 2: MLN8237 50 mg- Breast Cancer | Phase 2: MLN8237 50 mg- Gastric Cancer | Phase 2: MLN8237 50 mg- HNSCC | Phase 2: MLN8237 50 mg- NSCLC | Phase 2: MLN8237 50 mg- SCLC
Number analyzed (Participants) | 9 | 4 | 4 | 1 | 10
days | 169 [85 to 313] | 198 [146 to 501] | 79 [46 to 95] | NA [NA to NA] — Median and 95% confidence interval were not estimable because the single participant in this group was censored. | 125 [93 to 365]

6. Secondary Outcome: Phase 2: Number of Participants Reporting One or More Treatment-emergent Adverse Events and Serious Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; or congenital anomaly; or a medically important event.
Time Frame: Baseline up to 30 days after the last dose of study drug
Population: Safety population included all participants who received any amount of alisertib.
Measure: Number; unit: participants
Arm/Group | Phase 2: MLN8237 50 mg- Breast Cancer | Phase 2: MLN8237 50 mg- Gastric Cancer | Phase 2: MLN8237 50 mg- HNSCC | Phase 2: MLN8237 50 mg- NSCLC | Phase 2: MLN8237 50 mg- SCLC
Number analyzed (Participants) | 53 | 55 | 55 | 26 | 60
participants
  Adverse Events | 52 | 52 | 54 | 26 | 57
  Serious Adverse Events | 23 | 30 | 19 | 8 | 28

7. Secondary Outcome: Phase 1: Cmax- Maximum Observed Plasma Concentration for Alisertib
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Days 1 and 7: predose, 30 minutes, 1, 2, 3, 4, 6, 8, and 12 hours post-dose
Population: Pharmacokinetic (PK)-Evaluable population included all participants who had sufficient dosing data and alisertib concentration-time data to permit calculation of alisertib PK parameters in Phase 1 where Days 1 and 7 assessment were available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole (nM)
Groups:
- Phase 1: MLN8237 50 mg (Including Pancreatic Cancer): MLN8237 (alisertib) 50 mg, enteric-coated tablets, orally, twice daily for 7 days followed by 14 days of rest period in 21-day treatment cycles for a maximum of 24 months, or until progressive disease, unacceptable treatment-related toxicity, or initiation of a different anticancer therapy during Phase 1 portion of the study. Included participants from dose-escalation cohort or pancreatic cancer cohort who received alisertib 50 mg twice daily.
Arm/Group | Phase 1: MLN8237 10 mg | Phase 1: MLN8237 20 mg | Phase 1: MLN8237 40 mg | Phase 1: MLN8237 50 mg (Including Pancreatic Cancer) | Phase 1: MLN8237 60 mg
Number analyzed (Participants) | 1 | 3 | 4 | 13 | 3
nanomole (nM)
  Day 1 (n = 1, 3, 4, 13, 3) | 297 | 602 (15) | 949 (49) | 1619 (39) | 1696 (37)
  Day 7 (n = 1, 3, 3, 12, 2) | 981 | 1279 (35) | 1830 (39) | 2907 (49) | 3027 (NA) — A minimum of 2 patients are required to show the mean and geometric mean, and at least 3 patients are required to show the standard deviation and CV. CV = std/mean*100

8. Secondary Outcome: Phase 1: Tmax- Time to Reach the Maximum Plasma Concentration (Cmax) for Alisertib
Description: Tmax: Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax.
Time Frame: Days 1 and 7: predose, 30 minutes, 1, 2, 3, 4, 6, 8, and 12 hours postdose
Population: PK-Evaluable population included all participants who had sufficient dosing data and alisertib concentration-time data to permit calculation of alisertib PK parameters in Phase 1 where Day 1 and Day 7 assessment were available.
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1: MLN8237 10 mg | Phase 1: MLN8237 20 mg | Phase 1: MLN8237 40 mg | Phase 1: MLN8237 50 mg (Including Pancreatic Cancer) | Phase 1: MLN8237 60 mg
Number analyzed (Participants) | 1 | 3 | 4 | 13 | 3
hours
  Day 1 (n = 1, 3, 4, 13, 3) | 2.9 | 2.0 [2 to 2.9] | 3.2 [2.8 to 6] | 2.2 [1.7 to 11] | 6.0 [3 to 7.9]
  Day 7 (n = 1, 3, 3, 12, 2) | 3.1 | 3.0 [1 to 6] | 3.0 [2 to 6] | 2.4 [0 to 8] | 2.8 [2.6 to 3.0]

9. Secondary Outcome: Phase 1: AUC(0-tau): Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval for Alisertib
Description: Area under the plasma concentration-time curve during a dosing interval, where tau is the length of the dosing interval.
Time Frame: Days 1 and 7: predose, 30 minutes, 1, 2, 3, 4, 6, 8, and 12 hours postdose
Population: PK-Evaluable population included all participants who had sufficient dosing data and alisertib concentration-time data to permit calculation of alisertib PK parameters in Phase 1 where Days 1 and 7 assessment were available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole*hour (nM*hr)
Arm/Group | Phase 1: MLN8237 10 mg | Phase 1: MLN8237 20 mg | Phase 1: MLN8237 40 mg | Phase 1: MLN8237 50 mg (Including Pancreatic Cancer) | Phase 1: MLN8237 60 mg
Number analyzed (Participants) | 1 | 3 | 4 | 13 | 3
nanomole*hour (nM*hr)
  Day 1 (n = 1, 3, 4, 13, 3) | 2640 | 3495 (19) | 5015 (57) | 10736 (48) | 13932 (42)
  Day 7 (n = 1, 3, 3, 11, 2) | 8660 | 10184 (24) | 13694 (59) | 20867 (49) | 28709 (NA) — A minimum of 2 patients are required to show the mean and geometric mean, and at least 3 patients are required to show the standard deviation and CV. CV = std/mean*100

10. Secondary Outcome: Phase 1: Terminal Phase Elimination Half-life (T1/2) for Alisertib
Description: Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Time Frame: Day 7: predose, 30 minutes, 1, 2, 3, 4, 6, 8, and 12 hours postdose
Population: PK-Evaluable population included all participants who had sufficient dosing data and alisertib concentration-time data to permit calculation of alisertib PK parameters in Phase 1 where Day 7 assessment was available.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Phase 1: MLN8237 10 mg | Phase 1: MLN8237 20 mg | Phase 1: MLN8237 40 mg | Phase 1: MLN8237 50 mg (Including Pancreatic Cancer) | Phase 1: MLN8237 60 mg
Number analyzed (Participants) | 1 | 3 | 2 | 9 | 2
hours | 20.6 | 16.0 (1.2) | 19.0 (NA) — A minimum of 2 patients are required to show the mean and geometric mean, and at least 3 patients are required to show the standard deviation and CV. CV = std/mean*100 | 20.8 (10.3) | 27.8 (NA) — A minimum of 2 patients are required to show the mean and geometric mean, and at least 3 patients are required to show the standard deviation and CV. CV = std/mean*100

11. Secondary Outcome: Phase 1: Rac- Accumulation Ratio for Alisertib
Description: Rac was estimated as a ratio of AUC (0-tau) at Day 7 and AUC (0-tau) at Day 1. Area under the plasma concentration-time curve during a dosing interval, where tau is the length of the dosing interval.
Time Frame: Days 1 and 7: predose, 30 minutes, 1, 2, 3, 4, 6, 8, and 12 hours postdose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Phase 1: MLN8237 10 mg | Phase 1: MLN8237 20 mg | Phase 1: MLN8237 40 mg | Phase 1: MLN8237 50 mg (Including Pancreatic Cancer) | Phase 1: MLN8237 60 mg
Number analyzed (Participants) | 1 | 3 | 3 | 11 | 2
ratio | 3.3 | 3.0 (1.0) | 2.3 (0.4) | 2.2 (0.9) | 2.4 (NA) — A minimum of 2 patients are required to show the mean and geometric mean, and at least 3 patients are required to show the standard deviation and CV. CV = std/mean*100

12. Secondary Outcome: Phase 1: Peak to Trough Ratio for Alisertib
Description: Peak to trough ratio was estimated as a ratio of Cmax at Day 7 and the minimum observed plasma concentration (Ctrough) of alisertib at Day 7. Cmax is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve. Ctrough is the minimum plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Day 7: predose, 30 minutes, 1, 2, 3, 4, 6, 8, and 12 hours postdose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Phase 1: MLN8237 10 mg | Phase 1: MLN8237 20 mg | Phase 1: MLN8237 40 mg | Phase 1: MLN8237 50 mg (Including Pancreatic Cancer) | Phase 1: MLN8237 60 mg
Number analyzed (Participants) | 1 | 3 | 3 | 11 | 2
ratio | 1.7 | 2.1 (0.7) | 2.3 (1.4) | 2.3 (0.8) | 1.8 (NA) — A minimum of 2 patients are required to show the mean and geometric mean, and at least 3 patients are required to show the standard deviation and CV. CV = std/mean*100

13. Secondary Outcome: Phase 1: Steady State Oral Clearance (CLss/F) for Alisertib
Description: CL/F is apparent clearance of the drug from the plasma, calculated as the drug dose divided AUC(0-tau), expressed in liter per hour (L/hr).
Time Frame: Day 7: predose, 30 minutes, 1, 2, 3, 4, 6, 8, and 12 hours postdose
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Phase 1: MLN8237 10 mg | Phase 1: MLN8237 20 mg | Phase 1: MLN8237 40 mg | Phase 1: MLN8237 50 mg (Including Pancreatic Cancer) | Phase 1: MLN8237 60 mg
Number analyzed (Participants) | 1 | 3 | 3 | 11 | 2
L/hr | 2.2 | 3.8 (22) | 5.6 (72) | 4.6 (39) | 4.0 (NA) — A minimum of 2 patients are required to show the mean and geometric mean, and at least 3 patients are required to show the standard deviation and CV. CV = std/mean*100

14. Secondary Outcome: Phase 2: Relationship Between Clinical Response and Molecular Markers of Response
Description: In SCLC,chemo-sensitive/resistant population were analyzed;in breast cancers,ER2 and ER2 status were analyzed.HR+ =estrogen receptor-positive or progesterone receptor-positive. HER+ =human epidermal growth factor receptor 2 (HER2). Triple negative =negative for estrogen receptors, progesterone receptors, and HER2.Clinical response according to RECIST version 1.1. CR:complete disappearance of all target lesions,non-target disease,except nodal disease;all nodes decrease to normal (short axis <10 mm);no new lesions. PR:>=30% decrease under baseline of the sum of diameters of all target lesions (SLD);short axis was used in the sum for target nodes,longest diameter used in the sum for all other target lesions;no unequivocal progression of non-target disease;no new lesions. Progressive Disease (PD): >=20% rise in SLD from the smallest value on study;unequivocal progression of existing non-target lesions. Stable Disease (SD):Neither sufficient shrinkage for PR nor sufficient increase for PD.
Time Frame: 12 months
Population: Response-Evaluable population. Data is reported only for SCLC and breast cancer cohorts becuase these cohorts showed clinical meaningful single agent activity, thus subgroup analysis were done to assess whether a particular subgroup of participants was more or less responsive to alisertib. Rest of the cohorts did not show meaningful activity.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: MLN8237 50 mg- Breast Cancer | Phase 2: MLN8237 50 mg- Gastric Cancer | Phase 2: MLN8237 50 mg- HNSCC | Phase 2: MLN8237 50 mg- NSCLC | Phase 2: MLN8237 50 mg- SCLC
Number analyzed (Participants) | 49 | 0 | 0 | 0 | 48
percentage of participants
  HR+: CR (n=26, 0, 0, 0, 0) | 0 [NA to NA] — Confidence interval was not calculated since none of the participants had the event in this category. |  |  |  | NA [NA to NA] — HER2 or ER2 analysis was not analyzed for SCLC cohort as per planned analysis.
  HR+: PR (n=26, 0, 0, 0, 0) | 23 [9 to 44] |  |  |  | NA [NA to NA] — HER2 or ER2 analysis was not analyzed for SCLC cohort as per planned analysis.
  HR+: SD (n=26, 0, 0, 0, 0) | 65 [44 to 83] |  |  |  | NA [NA to NA] — HER2 or ER2 analysis was not analyzed for SCLC cohort as per planned analysis.
  HR+: PD (n=26, 0, 0, 0, 0) | 12 [2 to 30] |  |  |  | NA [NA to NA] — HER2 or ER2 analysis was not analyzed for SCLC cohort as per planned analysis.
  HER+: CR (n=9, 0, 0, 0, 0) | 0 [NA to NA] — Confidence interval was not calculated since none of the participants had the event in this category. |  |  |  | NA [NA to NA] — HER2 or ER2 analysis was not analyzed for SCLC cohort as per planned analysis.
  HER+: PR (n=9, 0, 0, 0, 0) | 22 [3 to 60] |  |  |  | NA [NA to NA] — HER2 or ER2 analysis was not analyzed for SCLC cohort as per planned analysis.
  HER+: SD (n=9, 0, 0, 0, 0) | 36 [13 to 65] |  |  |  | NA [NA to NA] — HER2 or ER2 analysis was not analyzed for SCLC cohort as per planned analysis.
  HER+: PD (n=9, 0, 0, 0, 0) | 44 [14 to 79] |  |  |  | NA [NA to NA] — HER2 or ER2 analysis was not analyzed for SCLC cohort as per planned analysis.
  Triple Negative: CR (n=14, 0, 0, 0, 0) | 0 [NA to NA] — Confidence interval was not calculated since none of the participants had the event in this category. |  |  |  | NA [NA to NA] — HER2 or ER2 analysis was not analyzed for SCLC cohort as per planned analysis.
  Triple Negative: PR (n=14, 0, 0, 0, 0) | 7 [0 to 34] |  |  |  | NA [NA to NA] — HER2 or ER2 analysis was not analyzed for SCLC cohort as per planned analysis.
  Triple Negative: SD (n=14, 0, 0, 0, 0) | 36 [13 to 65] |  |  |  | NA [NA to NA] — HER2 or ER2 analysis was not analyzed for SCLC cohort as per planned analysis.
  Triple Negative: PD (n=14, 0, 0, 0, 0) | 57 [29 to 82] |  |  |  | NA [NA to NA] — HER2 or ER2 analysis was not analyzed for SCLC cohort as per planned analysis.
  Chemotherapy Refractory:CR(n=0,0,0,0,12) | NA [NA to NA] — Chemo-sensitive or resistent analysis was not analyzed for breast cancer cohort as per planned analysis. |  |  |  | 0 [NA to NA] — Confidence interval was not calculated since none of the participants had the event in this category.
  Chemotherapy Refractory:PR(n=0,0,0,0,12) | NA [NA to NA] — Chemo-sensitive or resistent analysis was not analyzed for breast cancer cohort as per planned analysis. |  |  |  | 25 [5 to 57]
  Chemotherapy Refractory:SD(n=0,0,0,0,12) | NA [NA to NA] — Chemo-sensitive or resistent analysis was not analyzed for breast cancer cohort as per planned analysis. |  |  |  | 25 [5 to 57]
  Chemotherapy Refractory:PD(n=0,0,0,0,12) | NA [NA to NA] — Chemo-sensitive or resistent analysis was not analyzed for breast cancer cohort as per planned analysis. |  |  |  | 50 [21 to 79]
  Chemotherapy Sensitive: CR(n=0,0,0,0,36) | NA [NA to NA] — Chemo-sensitive or resistent analysis was not analyzed for breast cancer cohort as per planned analysis. |  |  |  | 0 [NA to NA] — Confidence interval was not calculated since none of the participants had the event in this category.
  Chemotherapy Sensitive: PR(n=0,0,0,0,36) | NA [NA to NA] — Chemo-sensitive or resistent analysis was not analyzed for breast cancer cohort as per planned analysis. |  |  |  | 19 [8 to 36]
  Chemotherapy Sensitive: SD(n=0,0,0,0,36) | NA [NA to NA] — Chemo-sensitive or resistent analysis was not analyzed for breast cancer cohort as per planned analysis. |  |  |  | 36 [21 to 54]
  Chemotherapy Sensitive: PD(n=0,0,0,0,36) | NA [NA to NA] — Chemo-sensitive or resistent analysis was not analyzed for breast cancer cohort as per planned analysis. |  |  |  | 44 [28 to 62]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days after the last dose of study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Phase 1: MLN8237- Dose Escalation: MLN8237 (alisertib) 10, 20, 30, 40, 50, or 60 mg enteric-coated tablets, orally, twice daily, for 7 days followed by 14 days of rest period in 21-day treatment cycles for a maximum of 24 months, or until progressive disease, unacceptable treatment-related toxicity, or initiation of a different anticancer therapy in participants enrolled in dose escalation cohort during Phase 1 portion of the study.
Arm/Group | Phase 1: MLN8237- Dose Escalation | Phase 1: MLN8237 50 mg- Pancreatic Cancer | Phase 2: MLN8237 50 mg- Breast Cancer | Phase 2: MLN8237 50 mg- Gastric Cancer | Phase 2: MLN8237 50 mg- HNSCC | Phase 2: MLN8237 50 mg- NSCLC | Phase 2: MLN8237 50 mg- SCLC
Serious Adverse Events (participants affected / at risk) | 13/23 | 1/1 | 23/53 | 30/55 | 19/55 | 8/26 | 28/60
Other Adverse Events (participants affected / at risk) | 23/23 | 1/1 | 52/53 | 52/55 | 54/55 | 26/26 | 55/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: MLN8237- Dose Escalation (N=23) | Phase 1: MLN8237 50 mg- Pancreatic Cancer (N=1) | Phase 2: MLN8237 50 mg- Breast Cancer (N=53) | Phase 2: MLN8237 50 mg- Gastric Cancer (N=55) | Phase 2: MLN8237 50 mg- HNSCC (N=55) | Phase 2: MLN8237 50 mg- NSCLC (N=26) | Phase 2: MLN8237 50 mg- SCLC (N=60)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 4 | 1 | 3 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 2 | 2 | 2 | 0 | 4
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 2 | 2 | 1 | 0 | 2
Asthenia (General disorders) | 1 | 0 | 2 | 2 | 1 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 2 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 3 | 0 | 1 | 1 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 1 | 2 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 2
Sepsis (Infections and infestations) | 0 | 0 | 3 | 0 | 1 | 0 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 4
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arterial injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhagic ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: MLN8237- Dose Escalation (N=23) | Phase 1: MLN8237 50 mg- Pancreatic Cancer (N=1) | Phase 2: MLN8237 50 mg- Breast Cancer (N=53) | Phase 2: MLN8237 50 mg- Gastric Cancer (N=55) | Phase 2: MLN8237 50 mg- HNSCC (N=55) | Phase 2: MLN8237 50 mg- NSCLC (N=26) | Phase 2: MLN8237 50 mg- SCLC (N=60)
Fatigue (General disorders) | 13 | 1 | 29 | 24 | 26 | 15 | 27
Neutropenia (Blood and lymphatic system disorders) | 10 | 0 | 31 | 23 | 25 | 15 | 21
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 0 | 26 | 21 | 24 | 11 | 16
Anaemia (Blood and lymphatic system disorders) | 4 | 1 | 20 | 25 | 24 | 13 | 16
Diarrhoea (Gastrointestinal disorders) | 10 | 0 | 27 | 21 | 15 | 9 | 17
Nausea (Gastrointestinal disorders) | 11 | 0 | 15 | 18 | 14 | 12 | 18
Decreased appetite (Metabolism and nutrition disorders) | 13 | 0 | 13 | 15 | 12 | 5 | 18
Stomatitis (Gastrointestinal disorders) | 9 | 0 | 24 | 11 | 14 | 4 | 12
Vomiting (Gastrointestinal disorders) | 8 | 1 | 11 | 16 | 13 | 6 | 10
Leukopenia (Blood and lymphatic system disorders) | 8 | 0 | 18 | 8 | 14 | 7 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1 | 11 | 14 | 7 | 6 | 11
Somnolence (Nervous system disorders) | 0 | 0 | 15 | 8 | 11 | 3 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 11 | 9 | 9 | 3 | 9
Constipation (Gastrointestinal disorders) | 2 | 0 | 9 | 11 | 9 | 5 | 5
Pyrexia (General disorders) | 3 | 0 | 5 | 13 | 11 | 3 | 4
Headache (Nervous system disorders) | 2 | 0 | 11 | 1 | 6 | 4 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 9 | 1 | 10 | 3 | 5
Oedema peripheral (General disorders) | 3 | 0 | 9 | 11 | 2 | 3 | 4
Insomnia (Psychiatric disorders) | 1 | 0 | 6 | 7 | 6 | 3 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 7 | 6 | 4 | 3 | 5
White blood cell count decreased (Investigations) | 3 | 0 | 5 | 4 | 4 | 1 | 10
Dehydration (Metabolism and nutrition disorders) | 6 | 0 | 7 | 3 | 2 | 3 | 4
Dizziness (Nervous system disorders) | 2 | 0 | 3 | 2 | 6 | 5 | 7
Weight decreased (Investigations) | 3 | 0 | 5 | 2 | 6 | 2 | 5
Abdominal pain (Gastrointestinal disorders) | 4 | 0 | 9 | 3 | 3 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 4 | 4 | 4 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 6 | 6 | 2 | 1 | 7
Asthenia (General disorders) | 0 | 0 | 3 | 4 | 5 | 3 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 5 | 4 | 2 | 2 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 2 | 4 | 2 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4 | 0 | 5 | 3 | 3
Oral candidiasis (Infections and infestations) | 5 | 0 | 5 | 2 | 3 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 2 | 6 | 1 | 1 | 3
Confusional state (Psychiatric disorders) | 2 | 0 | 3 | 1 | 2 | 1 | 6
Anxiety (Psychiatric disorders) | 1 | 0 | 3 | 5 | 2 | 0 | 3
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 4 | 6 | 3 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 1 | 1 | 2 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 2 | 2 | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review in advance of publication.